CLINICAL TRIAL: NCT06048029
Title: Laparoscopic Cholecystectomy in Children. Risk Factors for Conversion. A Prospective Study .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Korashy, primary investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cholecystectomy
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Laparoscopic Cholecystectomy in Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Cholecystectomy in children (Other): Evaluate preoperative and operative risk factors for laparoscopic cholecystectomy compared to open cholecystetcomy
  Interventions: Procedure: laparscopic Cholecystectomy in children
- Open Cholecystectomy in children (Other): Evaluate preoperative and operative risk factors for open cholecystectomy compared to laparoscopic cholecystetcomy
  Interventions: Procedure: laparscopic Cholecystectomy in children

INTERVENTIONS:
Procedure: laparscopic Cholecystectomy in children — Evaluate preoperative and operative risk factors for conversion of laparoscopic cholecystectomy to open cholecystectomy
  Other Names: open Cholecystectomy in children

SUMMARY:
Cholecystectomy is the most common procedure in biliary surgery which may be open or laparoscopic.laparoscopic cholecystectomy is widely accepted as the gold standard technique in both adults and children .over recent years there has been a significant increase in paediatric cholecystectomies alongside a rising incidence of childhood gall stones.

DETAILED DESCRIPTION:
The majority of paediatric gallstones are related to haemolytic diseases such as hereditary spherocytosis. In recent decades, the incidence of gallstone disease in children has risen which may be related to the epidemic of paediatric obesity and improved survival of critically ill neonates who have received long-term total parenteral nutrition or correction of abnormalities resulting in increased incidence of cholelithiasis in the paediatric population such as short gut syndrome.The rate of conversion to open cholecystectomy ranges between 2% and 20%. Certain preoperative and operative factors can reliably predict the chances of conversion to the open procedure. Until recently large studies are lacking of assessment of the risk factors that my be responsible for conversion of laparoscopic cholecystectomy to open cholecystectomy . This study aims to assess preoperative and operative risk factors for conversion to open surgery .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age less than 18 years old presented to assiut university hospitals at pediatric surgeey unit.
2. fit for surgery

Exclusion Criteria:

1. patients with co-existent common bile duct stones based on imaging and biochemical criteria.
2. Patients with Pancreatitis .
3. Patients with previous upper abdominal surgery.

5_Significant medical disease rendering patient unfit for Laparoscopic surgery (e.g. Chronic Pulmonary Disease, significant Cardiac Disease)

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-03 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Cholecystectomy in children | one year
  Evaluate and the risk factors for conversion of laparoscopic to open cholecystectomy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gadacz TR. Update on laparoscopic cholecystectomy, including a clinical pathway. Surg Clin North Am. 2000 Aug;80(4):1127-49. doi: 10.1016/s0039-6109(05)70217-6. PMID 10987028
- [Background] van der Steeg HJ, Alexander S, Houterman S, Slooter GD, Roumen RM. Risk factors for conversion during laparoscopic cholecystectomy - experiences from a general teaching hospital. Scand J Surg. 2011;100(3):169-73. doi: 10.1177/145749691110000306. PMID 22108744
- [Background] Rothstein DH, Harmon CM. Gallbladder disease in children. Semin Pediatr Surg. 2016 Aug;25(4):225-31. doi: 10.1053/j.sempedsurg.2016.05.005. Epub 2016 May 11. PMID 27521713
- [Background] Khoo AK, Cartwright R, Berry S, Davenport M. Cholecystectomy in English children: evidence of an epidemic (1997-2012). J Pediatr Surg. 2014 Feb;49(2):284-8; discussion 288. doi: 10.1016/j.jpedsurg.2013.11.053. Epub 2013 Nov 18. PMID 24528968
- [Background] Zeidan MM, Pandian TK, Ibrahim KA, Moir CR, Ishitani MB, Zarroug AE. Laparoscopic cholecystectomy in the pediatric population: a single-center experience. Surg Laparosc Endosc Percutan Tech. 2014 Jun;24(3):248-50. doi: 10.1097/SLE.0b013e3182a4c039. PMID 24887542
- [Background] Palser TR, Ceney A, Navarro A, Swift S, Bowrey DJ, Beckingham IJ. Variation in laparoscopic anti-reflux surgery across England: a 5-year review. Surg Endosc. 2018 Jul;32(7):3208-3214. doi: 10.1007/s00464-018-6038-y. Epub 2018 Jan 24. PMID 29368285
- [Background] Padbury RTA. Day-only laparoscopic cholecystectomy in 2021. ANZ J Surg. 2021 Apr;91(4):484. doi: 10.1111/ans.16686. No abstract available. PMID 33847061
- [Background] Rio-Tinto R, Canena J. Endoscopic Treatment of Post-Cholecystectomy Biliary Leaks. GE Port J Gastroenterol. 2021 Jul;28(4):265-273. doi: 10.1159/000511527. Epub 2020 Dec 8. PMID 34386554